CLINICAL TRIAL: NCT04429711
Title: Ivermectin vs. Placebo for the Treatment of Patients With Mild to Moderate COVID-19 to Prevent Progression to Severe Infection and to Decrease Viral Shedding - A Double Blind , Randomized Controlled Trial
Brief Title: Ivermectin vs. Placebo for the Treatment of Patients With Mild to Moderate COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Eli Schwartz MD, DTMH, Prinicipal Investigator, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-20-7156-ES-CTIL
Record Dates: First submitted 2020-05-24; First posted 2020-06-12 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Double blind randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVERMECTIN (Placebo Comparator)
  Interventions: Drug: Ivermectin Oral Product
- PLACEBO (Active Comparator)
  Interventions: Drug: Ivermectin Oral Product

INTERVENTIONS:
Drug: Ivermectin Oral Product — 3mg Capsules, 12-15mg/ day for 3 days

SUMMARY:
Ivermectin which is an FDA-approved broad spectrum anti-parasitic agent, has also anti-viral activity. In vitro study have shown its activity against SARS-CoV-2, however its clinical effect on patients with COVID-19 never been tested.

In this RCT we would like to evaluate the effect of Ivermectin on reduction of viral shedding among mild to moderate COVID-19 patients, and in shortening the symptom resolution time.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion will include non-pregnant adult (>18 years old) with molecular confirmation of COVID-19. [Participants will be eligible in a period of no longer than 72 hours after exposure].

Exclusion Criteria:

* Severe infection ( defined as need for invasive or non-invasive ventilator support, ECMO or shock requiring vasopressor support).
* Weight below 40Kg or above 100Kg
* Unable to take oral medication
* Known allergy to the drugs
* Pregnancy or breast feeding
* Participating in another RCT for treatment of COVID-19.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Viral clearance at day 6 | Outcome will be determined till 6 days post intervention
  The primary outcome will be the viral clearance at day 6 in the intervention group compared to placebo.
Viral shedding duration | Outcome will be determined till 14 days post intervention
  Secondary outcomes: viral shedding duration (time between first positive PCR to last of two consecutive negative tests)
Symptoms clearance time | Outcome will be determined till 14 days post intervention
  Time between drug treatment and symptoms resolution

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel